CLINICAL TRIAL: NCT06548997
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GZR18 Injection in Healthy Subjects Following Single Dose and Once-weekly Dose for 2 Consecutive Weeks Until Reaching the Target Dose
Brief Title: A Phase I Study of GZR18 Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLP-CH1002
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GZR18 (Experimental)
  Interventions: Drug: GZR18
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR18 — 5 μg/kg-maximum tolerated dose (MTD), single dose or two doses
  Arms: GZR18
Other: Placebo — administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
This trial is conducted in China. The aim of the trial is to evaluate the safety and tolerability of GZR18 injection in healthy subjects following single dose and once-weekly dose for 2 consecutive weeks until reaching the target dose.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects sign informed consent voluntarily.
* 2. Chinese adult subjects, male or female.
* 3. Age 18-55 at screening (both included).
* 4. At screening and baseline, 19.0 kg/m2 ≤ BMI ≤ 26.0 kg/m2 (male ≥55.0 kg, female ≥45.0 kg).
* 5. Female subjects were human chorionic gonadotophin (HCG) negative at screening and baseline.

Exclusion Criteria:

* 1. History of dizziness with blood and needles.
* 2. Known or suspected allergy to study related products; or a history of drug and food allergies; or a history of allergy-related diseases.
* 3. Participants who participated in other clinical trials and were given the investigational drug or medical device intervention within 90 days prior to screening.
* 4. Blood donation, surgery, or trauma with significant blood loss (more than or equal to 400 mL, except for menstrual blood loss in women) within 12 weeks prior to screening.
* 5. Any clinically significant medical history judged by the investigator, including but not limited to: lung, gastrointestinal, liver, nervous system, kidney, genitourinary and endocrine, skin, or blood disorders, especially a personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2 , and a history of pancreatitis (acute or chronic).
* 6. At screening or baseline, physical examination showed clinically significant abnormalities judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
TEAE | after 28/35 days of treatment
  Incidence of treatment-emergent adverse events (TEAE)

SECONDARY OUTCOMES:
Cmax | 28/35 days
  The peak concentration after reaching the target dose
AUClast | 28/35 days
  the area under the concentration-time curve from 0 to the last time that the concentration can be accurately measured
AUC0-inf | 28/35 days
  the area under the concentration-time curve from 0 to infinity
Tmax | 28/35 days
  the peak time
λz | 28/35 days
  the elimination rate constant
t1/2 | 28/35 days
  the half-life
tlag | 28/35 days
  retention time
CL/F | 28/35 days
  apparent clearance rate
Vz/F | 28/35 days
  apparent volume of distribution
AUC%extra | 28/35 days
  extrapolation percentage of AUC0-in
MRT | 28/35 days
  average retention time
AUCglucose0-14h | 28/35 days
  area under the concentration-time curve of fasting blood glucose from 0 to 14 hours after each administration
AUCc-peptide0-14h | 28/35 days
  area under the concentration-time curve of fasting C-peptide from 0 to 14 hours after each administration
AUCinsulin0-14h | 28/35 days
  area under the concentration-time curve of fasting insulin from 0 to 14 hours after each administration
body weight | 28/35 days
body mass index (BMI） | 28/35 days

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao, Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, China